CLINICAL TRIAL: NCT00745303
Title: Effect of Tai Chi Chuan on Autonomic Nervous Modulation, Blood Lipid and Cytokines Production in Aged Subjects
Brief Title: Effect of Tai Chi Chuan on Autonomic Nervous Modulation in Aged Subjects
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Cho-yu Chan, MD, Taipei Veterans General Hospital
Other Study IDs: VGH91-365-1
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Healthy Subjects
Keywords: Tai Chi Chuan; Lipid; Cytokine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample obtained from each subject was withdrawn for the quantitative measurements of total cholesterol (TC), high-density lipoprotein--cholesterol (HDL-C), high-density lipoprotein--cholesterol (LDL-C), triglyceride (TG), fasting blood sugar (FBS), and uric acid (UA). The immunoenzymometric assays for the quantitative measurement of tumor necrosis factor-α (TNF-α) and interferon-γ (IFN-γ) in the serum were also performed on the blood sample from each subject.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects in this group received TCC training for 3 months
  Interventions: Procedure: Tai Chi Cuan
- 2: Subjects in this group received no TCC training within 3 months

INTERVENTIONS:
Procedure: Tai Chi Cuan — Tai Chi Cuan training for 3 months
  Other Names: Yang's Tai Chi Cuan
  Groups: 1

SUMMARY:
Since Tai Chi Chuan (TCC) training has been shown to be beneficial to the cardiopulmonary function of the subject, TCC might have a beneficial effect on the pulmonary function, autonomic nervous modulation, lipid profile, and cytokines production in the aged subjects.

DETAILED DESCRIPTION:
Tai Chi Chuan (TCC) is a traditional Oriental conditioning exercise or calisthenics that is believed by many people around the world to be good for the health. The frequently claimed reason for this merit of TCC is that it can improve the cardiopulmonary function and immunity of the subject who practice it continuously. TCC has been shown to delay the decline of aerobic power, improve the cardiopulmonary function, balance and strength of the subjects. One study has demonstrated that TCC could reduce tension, anxiety, and mood disturbance. However, few studies have examined the effect of TCC on the blood lipid profile and immunity of the TCC practitioners. Another study reported that 12-week programme of regular TCC exercise enhanced functional mobility, personal health expectations, and regulatory T cell function. It has also been shown that an appropriate combination of TCC exercise program with diabetic medication might improve both glucose metabolism and immunity in type 2 diabetic patients. Since TCC training has been shown to be beneficial to the cardiopulmonary function of the subject, TCC may also have an effect on the blood lipid profile and immunity of the subjects. We hypothesize that TCC might have a beneficial effect on the pulmonary function, autonomic nervous modulation, lipid profile, and cytokines production in the aged subjects. Thus, the aim of this study was to examine whether or not TCC have these effects in the aged subjects.

ELIGIBILITY:
Inclusion Criteria:

* All subjects included in this study had normal lifestyles, and were capable of daily activities without limitations.

Exclusion Criteria:

* Subjects who had major cardiopulmonary disease or were on regular medicine for diabetes mellitus, hypertension, renal or liver disease were not included in the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy aged subjects
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2002-05; Primary Completion 2003-05 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
TCC training for 3 months can improve the pulmonary function, glucose availability and lipid profile, and increase the cytokines production and vagal modulation in aged subjects. | 3 months

SECONDARY OUTCOMES:
Other effects of TCC observed | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Deng Kuo, MD,PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Lu WA, Kuo CD. The effect of Tai Chi Chuan on the autonomic nervous modulation in older persons. Med Sci Sports Exerc. 2003 Dec;35(12):1972-6. doi: 10.1249/01.MSS.0000099242.10669.F7. PMID 14652490